CLINICAL TRIAL: NCT04671056
Title: A Single Center, Open-Label, Drug Interaction Study of MGL-3196 With Pioglitazone and to Assess Food Effect in Healthy Subjects
Brief Title: Drug Interaction Study of MGL-3196 With Pioglitazone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGL-3196-09
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Healthy
MeSH Terms: interventions — resmetirom; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MGL-3196 100 mg tablet plus Pioglitazone 15 mg tablet (Experimental): MGL-3196 administered orally plus Pioglitazone administered orally on 2 separate days
  Interventions: Drug: MGL-3196; Drug: Pioglitazone 15mg

INTERVENTIONS:
Drug: MGL-3196 — MGL-3196 100 mg tablet administered orally in the morning for 13 days
Drug: Pioglitazone 15mg — Pioglitazone 15 mg tablet administered orally on 2 separate days, initially on one day alone and again after MGL-3196 has been dosed to steady-state

SUMMARY:
The purpose of this study is to determine whether the single-dose pharmacokinetics (AUC) of pioglitazone are affected by chronic dosing with MGL-3196 100 mg/day in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing and able to provide written informed consent
* Healthy, non-smoking male or female between the ages of 19 and 55 years (inclusive)
* Body weight > 50 kg and BMI between 18 and 32 kg/m2 (inclusive)
* If female, is non-pregnant and non-lactating. For females of non-childbearing potential, must have undergone sterilization procedures (hysteroscopic sterilization, bilateral tubal ligation or bilateral salpingectomy, hysterectomy, bilateral oophorectomy) at least 6 months prior to first dosing. Or, is postmenopausal with amenorrhea for at least 1 year prior to first dosing as verified by follicle stimulating hormone (FSH) at screening
* If female of childbearing potential, must use acceptable non-hormonal birth control (surgical sterilization of the partner, physical barrier method for at least 30 days prior to first dosing in addition to spermicide from the time of screening throughout study completion, non-hormonal intrauterine device for at least 3 months prior to first dosing, total abstinence from sexual intercourse for at least at least 3 months prior to first dosing and throughout study completion)
* If male and non-vasectomized, must agree to use a condom with spermicide or abstain from sexual intercourse from the first dose of study drug until 14 days beyond the last dose of study drug. No restrictions required for vasectomized male provided his vasectomy has been performed 3 months or more prior to Day 1. A male who has been vasectomized less than 3 months prior to study start must follow the same procedure as a non-vasectomized male.

Exclusion Criteria:

* Any clinically significant abnormal findings on physical examination, clinical laboratory tests or 12-lead ECG.
* Evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, renal, hepatic, neurological or psychiatric disease.
* Current or recent (<6 months) hepatobiliary disease; or AST, ALT or direct bilirubin greater than the upper limit of reference range at screening. Repeat testing is allowed per site standard procedures.
* Gilbert's syndrome.
* Pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function that could interfere with the absorption, metabolism, and/or excretion of study drug (Cholecystectomy is allowed).
* Abnormal screening ECG: including machine-read QTcF >450 msec in men and QTcF > 470 msec in women (confirmed by manual over read) or any rhythm other than normal sinus rhythm which is interpreted by the Investigator to be clinically significant.
* History of sensitivity to a similar study drug, thyroid medication, or a history of important drug or other allergy (except for untreated, asymptomatic seasonal allergies at time of dosing) unless deemed not clinically significant by the Investigator.
* Participation in another clinical trial of an investigational drug (or medical device) within the last 30 days prior to the Day 1, or who have been exposed to more than four new chemical entities within 12 months prior to Day 1.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
AUC from the time of dosing of pioglitazone as affected by chronic dosing with MGL-3196 100 mg/day in healthy subjects | 17 days

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No